CLINICAL TRIAL: NCT00589784
Title: Phase II Trial of Sunitinib (SU011248) in Patients With Recurrent or Inoperable Meningioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); University of Virginia (Other); University of Pittsburgh (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-135; NCT00561665 (obsolete NCT alias)
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: CNS Cancer; Meningioma; Intracranial Hemangiopericytoma; Hemangioblastoma; Neurofibromatosis
Keywords: Sunitinib; Brain Cancer; CNS Cancer; meningioma; intracranial hemangiopericytoma; hemangioblastoma; malignant meningioma; neurofibromatosis; neurofibromatosis type 1; neurofibromatosis type 2; 07-135
MeSH Terms: conditions — Central Nervous System Neoplasms; Meningioma; Hemangioblastoma; Neurofibromatoses; Brain Neoplasms; Neurofibromatosis 1; Neurofibromatosis 2 | interventions — Sunitinib

ARMS (1):
- Treatment (Experimental): Sunitinib will be administered at a dose of 50 mg orally once daily for four consecutive weeks, followed by a two-week rest period. Intra-patient dose reduction may be required depending on the type and severity of individual toxicity encountered. Imaging studies will be performed after every other cycle. Patients may continue on study as long as they are tolerating treatment and in the absence of disease progression.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — The study drug will be administered on an outpatient basis. The starting dose will be 50 mg daily for 28 days (4 consecutive weeks) followed by 14 days off for patients not on CYP3A4 inducers or inhibitors. A cycle equals 42 days.
  Other Names: Patients on strong CYP3A4 inducers should start at a dose of 62.5 mg and those; on strong CYP3A4 inhibitors should start at a dose of 37.5 mg. The dose should; be taken once daily at approximately the same time each day.; Patients are required to have a drug rest period of at least 14 days after; each dosing period. The start of the next cycle may be delayed if additional; time is required for the patient to recover from sunitinib-associated toxicity; experienced during the previous cycle. An interruption in therapy of greater; than 28 days must be approved by the PI. Dosing can be modified after; discussion with the study investigator. The study investigator may implement; dose suspension or reduction in order to ensure patient safety. Patients will; be given a diary to take home to record their sunitinib dosing.; This will be brought back to the clinic following each cycle of treatment.; SU011248

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, sunitinib has on patients and their tumors. At this time, no drugs are routinely used to treat meningioma, hemangioblastoma or hemangiopericytoma. Only surgery and radiation therapy are known to be useful.

Sunitinib is a drug approved for advanced kidney cancer. Sunitinib is also being studied for other tumors. It may be useful in the treatment of brain tumors because it can prevent formation of new blood vessels that allow tumor cells to survive and grow.

DETAILED DESCRIPTION:
This is a phase II study of Sunitinib in patients with recurrent or inoperable meningiomas. An exploratory study will be performed for patients with recurrent hemangiopericytoma or hemangioblastoma. There will be approximately 50 patients enrolled on this study (40 meningiomas and 10 hemangiopericytomas/hemangioblastomas). The treatment plan is to use daily SU11248 at a dose of 50 mg, using the established schedule of 4 weeks of treatment followed by two weeks of rest period, forming a six-week treatment cycle. A medical professional will see each patient at least every six weeks while on the medication for toxicity assessment and physical examination. Extent of disease evaluations will occur at baseline, two weeks, twelve weeks, 24 weeks, and every twelve weeks thereafter. These evaluations will include MRI of the brain (or CT head if a patient cannot undergo MRI) and MR perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven recurrent meningioma or intracranial hemangiopericytoma or hemangioblastoma. This includes benign, atypical, or malignant meningioma; patients with neurofibromatosis type 1 or 2 may participate.
* Patients with classic radiographic picture of meningioma may also enroll if not surgically accessible. In this instance the patient must be reviewed at multi-disciplinary brain tumor conference including neurosurgery and neuroradiology to determine that the patient is appropriate for this study.
* Unequivocal evidence for tumor progression by MRI (or CT scan if MRI is contraindicated). The scan must be performed within 14 days of registration.
* Steroids dosing - malignant meningiomas must be on stable dose for at least 5 days prior to baseline imaging. For patients with benign or atypical meningiomas, stable steroid doses are not required.
* Recent resection for recurrent tumor - patients will be eligible as long as they have recovered from the effects of surgery and have residual disease that can be evaluated. To best assess the extent of residual disease post-operatively, a CT/MRI should be done no later than 96 hours in the immediate post-operative period or at least 4 weeks post-operatively. If the 96 hour scan is more than 14 days before registration, it should be repeated. Because Sunitinib is a VEGF inhibitor that can carry many risks including thrombocytopenia, bleeding, hypertension, and stroke, patients must wait at least 14 days after surgery, without complication, before they may initiate study drug.
* Prior radiation therapy - patients may have been treated with standard external beam radiation, interstitial brachytherapy, or radiosurgery in any combination. An interval of ≥ 4 weeks (28 days) must have elapsed from the completion of radiation therapy to study entry and there must be subsequent evidence of tumor progression. Patients with prior interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based on PET, MR spectroscopy or surgical documentation of disease.
* Patients who have not had prior surgery or radiotherapy for their meningioma will be reviewed at multi-disciplinary brain tumor conference including neurosurgery and radiation oncology to determine that the patient is appropriate for this study.
* Prior therapy: There is no limitation on the number of prior surgeries, radiation therapy, radiosurgery treatments, or chemotherapy.
* All patients must sign an informed consent indicating that they are aware of the investigational nature of the study. Patients must sign an authorization for the release of their protected health information.
* Age ≥ 18 years old
* Karnofsky performance status ≥ 60%.
* ≥ 4 weeks since prior RT, stereotactic radiosurgery, or chemotherapy.
* Required Initial Laboratory Values (within 14 days of registration):

Absolute neutrophil count (ANC) ≥ 1,000/mm3

* Platelets ≥ 100,000/mm3
* hemoglobin ≥ 8gm/dl
* Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x local laboratory upper limit of normal (ULN)
* Creatinine ≤ 2.0 mg/dl
* PT, INR, and PTT ≤ 1.5 times institutional upper limits of normal
* Total serum bilirubin ≤ 1.5 - Patients with a history of NF may have other stable CNS tumors, such as schwannoma, acoustic neuroma, or ependymoma, but ONLY if these lesions have been stable in size for the preceding 6 months.

Exclusion Criteria:

* Patients with the history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix, unless in complete remission and off all therapy for the disease for a minimum of 3 years) are ineligible.
* Any prior TKI therapy (SU011248, Sorafenib, Semaxinib, Axitinib)
* Concomitant use of any other investigational drugs
* Concomitant use of enzyme-inducing anti-epileptic drugs.
* Concomitant use of St John's Wort.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias of NCI CTCAE Version 3.0 grade ≥ 2.
* Prolonged QTc interval on baseline EKG (>450 msec for males and >470 msec for females).
* Uncontrolled hypertension (>150/100 mm Hg despite optimal medical therapy). Patients are excluded if they have an elevated diastolic, an elevated systolic, or both.
* History of intracranial hemorrhage.
* Pre-existing thyroid abnormality, with thyroid function tests that cannot be maintained in the normal range with medication.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection.
* Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials, e.g. QOL, are allowed.
* Ongoing treatment with therapeutic doses of warfarin (low dose warfarin up to 2 mg daily for thromboembolic prophylaxis is allowed).
* Pregnancy or breast-feeding. Patients must be surgically sterile, postmenopausal, or agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate. Male patients must be surgically sterile or agree to use effective contraception. Women of childbearing potential must have a negative B-HCG pregnancy test documented within 14 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kaley, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Virginia Health Science Center, Charlottesville, Virginia

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Aggressive Memingioma: Patients with Aggressive Memingioma
- Exploratory Cohort: Patients with WHO grade I meningioma, HPC and hemangioblastoma
Period: Overall Study
Arm/Group | Aggressive Memingioma | Exploratory Cohort
Started | 36 | 14
Completed | 35 | 4
Not Completed | 1 | 10
Not completed — Withdrawal by Subject | 0 | 6
Not completed — Patient inevaluable | 1 | 0
Not completed — Adverse Event | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aggressive Memingioma | Exploratory Cohort | Total
Number analyzed (Participants) | 36 | 13 | 49
Age, Customized [Median (Full Range); unit: years]
  Median Age | 61 [27 to 85] | 48 [32 to 79] | 59 [27 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 22 | 8 | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: Determine the overall objective response
Time Frame: 1.5 years
Measure: Number; unit: participants
Arm/Group | Aggressive Memingioma | Exploratory Cohort
Number analyzed (Participants) | 35 | 4
participants
  Complete Response | 1 | 0
  Partial Response | 1 | 0
  Progression of Disease | 8 | 4
  Stable Disease | 25 | 0

ADVERSE EVENTS:
Groups:
- All Patients: All patients treated with Sunitinib (SU011248)
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 27/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=50)
CNS Hemorrhage (Nervous system disorders) | 4 (4)
Thrombic Microangiopathy (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Fatigue (General disorders) | 9 (9)
Thrombocytopenia (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5)
Lueukopenia (Blood and lymphatic system disorders) | 3 (3)
Hypertension (Cardiac disorders) | 4 (4)
Headache (General disorders) | 4 (4)
ALT (Blood and lymphatic system disorders) | 2 (2)
AST (Blood and lymphatic system disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Rash, Hand-Foot Reaction (Skin and subcutaneous tissue disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Prolonged QTc Interval (Cardiac disorders) | 1 (1)
Right Ventricular Enlargement (Cardiac disorders) | 1 (1)
Thrombosis/ Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperuricemia (Renal and urinary disorders) | 1 (1)
Gastrointestinal Perforation (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=50)
Leukopenia (Blood and lymphatic system disorders) | 31 (31)
Fatigue (General disorders) | 29 (29)
Thrombocytopenia (Respiratory, thoracic and mediastinal disorders) | 23 (23)
Diarrhea (Gastrointestinal disorders) | 22 (22)
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 (19)
AST (Blood and lymphatic system disorders) | 19 (19)
ALT (Blood and lymphatic system disorders) | 17 (17)
Nausea (Gastrointestinal disorders) | 17 (17)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (16)
Rash, Hand-Foot Reaction (Skin and subcutaneous tissue disorders) | 16 (16)
Mucositis (General disorders) | 13 (13)
Neutropenia (Blood and lymphatic system disorders) | 13 (13)
Dysgeusia (General disorders) | 13 (13)
Headache (General disorders) | 12 (12)
Vomiting (Gastrointestinal disorders) | 12 (12)
Hypertension (Cardiac disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes